CLINICAL TRIAL: NCT05667610
Title: Effect of an Immune-supportive Diet on Gut Permeability and Allergic Symptoms in Children With Peanut and/or Nut Allergy
Brief Title: Immune-supportive Diet and Gut Permeability in Allergic Children
Acronym: DIAMETER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Onze Lieve Vrouwe Gasthuis (Other)
Collaborators: Ekhaga foundation (Unknown); Rijnstate Hospital (Other); Noordwest Ziekenhuisgroep (Other); Erasmus Medical Center (Other); Wageningen University (Other); Amsterdam UMC (Other); Utrecht Institute for Pharmaceutical Sciences (Other); Diakonessenhuis, Utrecht (Other); Deventer Ziekenhuis (Other); Harvard University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL80586.100.22; W21.302 (Other: OLVG)
Record Dates: First submitted 2022-09-08; First posted 2022-12-28 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Peanut Allergy; Nut Allergy
Keywords: Gut permeability; Immune-supportive diet; Thresholds
MeSH Terms: conditions — Peanut Hypersensitivity; Nut Hypersensitivity | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Children in the intervention group will receive written and oral dietary advice by an allergy-specialist dietitian regarding their peanut or nut free diet according to standard care and, in addition, instructions on an individually tailored immune-supportive diet, including sample menus, recipes, shopping guide and product information.
  The dietitian will contact the patients every two to four-weeks as needed, either face-to-face, by video consult or using email or what app. Dietary compliance is orally checked by the dietitian, self-assessed dietary adherence and feasibility are score by Likert scale after 6 weeks and 3 months and dietary adherence is calculated by food diaries after 3 months. In addition, 22 healthy controls (without allergies),aged 4 to 12 years, will also be included.
Masking Description: The participants are randomly assigned to an intervention group or control group via castor.edc.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (immune-supportive diet) (Experimental): * Immune-supportive diet (for 4 months) on top of peanut and/or nut free diet. Foods are allocated into 3 food groups:
    1. Recommended in ample amounts: with an acknowledged beneficial role in immune health (first choice foods);
    2. Recommended in limited amounts: with an acknowledged beneficial role in immune health when used in limited amounts (second choice foods).
    3. Not recommended: with an acknowledged unfavourable role in immune health (third choice foods)
  * Self-assessed feasibility and adherence to the Immune-supportive diet (intervention group only) a by Likert scale after 2,5 and 4 months of dietary intervention;
  * Dietary adherence will be determined by the researchers after 4 months by calculating the number of first and second choice foods based on the food diaries after dietary intervention.
  Interventions: Other: Immune-supportive diet
- Control group (Active Comparator): - Peanut and/or nut free diet only
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Immune-supportive diet — The intervention includes a immune-supportive diet over a period of 4 months
  Arms: Intervention group (immune-supportive diet)
Other: Standard care — Standard care: Peanut or nut free diet
  Arms: Control group

SUMMARY:
Peanut and nut allergy can be life threatening. Some patients have very low threshold levels (i.e. the amounts of peanut and nuts to which the patients react), others react to higher doses. The reasons for these differences in threshold are not well understood. Patients with peanut and nut allergy often suffer from other allergic diseases (atopic dermatitis, hay fever and asthma). A disturbed gut microbiota composition and an increased gut permeability may explain the development of allergic disease. We hypothesize that increased gut permeability is related to low threshold levels to peanuts or nuts. In addition, as it is known that nutrition can influence our gut permeability, we also hypothesize that a healthful immune-supportive diet restores gut permeability and alleviates symptoms.

Therefore, the purpose of the study is to study in peanut and nut allergic children:

1. the relationship between gut permeability and threshold levels to peanut or nuts;
2. the effect of an immune-supportive diet on gut permeability, gut microbiome composition, coexisting allergic symptoms and quality of life

DETAILED DESCRIPTION:
The incidence of allergic asthma, atopic dermatitis and food allergy started to grow to epidemic proportions after the 1960s. Peanut and nut allergy are common food allergies. Peanut allergy affects 1.4 to 3.0% of the children. Peanut and nut allergy are often lifelong and may be severe. Peanut allergy is the leading cause of (fatal) food anaphylaxis. Once peanut and nut allergy have developed, there is currently no cure other than adhering to an avoidance diet and carrying and using intramuscular epinephrine or oral antihistamines in the case of accidental ingestion. Oral immunotherapy with peanut or nuts is only applied in research setting, however, it has several drawbacks and is still in its infancy.

Inter- and intra-individual differences in threshold in peanut allergy:

Threshold levels for peanut and nuts, the lowest amount of peanut or nuts causing a reaction, may largely vary between allergic children, for which there is no clear explanation. Thresholds can be determined during oral food challenge tests with peanut or nuts in the hospital. An international multi-center study found that 5% of the children react to a low threshold of 1.7 mg of peanut protein during the food challenge in the hospital, 7.4 mg of cashew nut protein and 0.29 mg of hazelnut protein during a food challenge in the hospital. These are only traces, while 50% react to 67 mg of peanut protein. This is around 1⁄3 of a peanut, thus also a small amount. These threshold levels demonstrate how careful patients have to be in their dietary behavior. Patients with a low threshold are very sensitive to peanut or nuts and are at greater risk to react to traces of allergenic protein which can be intentionally or unintentionally present in prepacked or unpacked food. Studies have shown that the lower the threshold, the greater the impact on the health-related quality of life of the child and their parents. It is poorly understood how these differences in sensitivity (threshold levels) between individuals can be explained. Sensitization to peanut or nuts, as demonstrated by levels specific immunoglobulin E (IgE) for peanut by blood testing or the size of the skin prick test with peanut or nuts cannot explain the difference in threshold level, because they have a low predictive value for the threshold. Infection diseases illness, exercise and sleep deprivation significantly reduce the threshold level in allergic adults. However, these co-factors are not relevant in all patients, specifically not in children, and cannot explain the large differences in threshold levels observed.

Peanut and nut allergy coincides with other atopic disease:

Peanut and nut allergic children frequently suffer from other food allergies, such as milk and egg, and other coexisting atopic (allergic) diseases such as atopic dermatitis, allergic rhinitis (hay fever) and allergic asthma, leading to a substantial allergic burden in children with peanut and nut allergy. Because of the burden of these allergic conditions, the quality of life of children with food allergy is decreased, however underestimated. and even lower compared to chronic diseases, e.g. lower than children with diabetes. All these coexisting allergic diseases are based on immunologic and chronic inflammatory processes. Asthma is a systemic inflammatory disorder with a close link between the upper and the lower airways. The majority of patients with asthma have concomitant rhinosinusitis. The respiratory system is also under the influence by co-morbid conditions related to the gastrointestinal tract (food sensitization, bowel inflammation), the skin (eczema, barrier dysfunction) as well as the nervous system (neuroimmunologic network, cognitive dysfunction).

Defective mucosal barrier function (leaky gut) or increased gut permeability as possible explanation for high prevalence of allergic disease and differences in threshold to peanut or nuts:

The steep increase of allergic diseases is attributed to several lifestyle changes due to urbanization and modernization, caesarean section, use of antibiotics, a westernized pro-inflammatory diet and obesity. Firstly, according to the generally accepted hypotheses, i.e. the hygiene hypothesis and the biodiversity hypothesis, all these changes lead to microbial dysbiosis and loss of microbial diversity in the gut, which are major reasons for inflammation, inappropriate immune responses and disease development, because there is a continuous crosstalk between the intestinal microbiome and our immune system through immunomodulatory signals. Allergic diseases, such as food allergy, asthma and atopic dermatitis are all characterized by a dysbiosis and reduced diversity of the microbiome.

Secondly, one of the most recent additional explanations for the increased prevalence of allergic disease is a defective epithelial (=mucosal) barrier in the skin, gut and lungs (the "extended epithelial barrier hypothesis"). Impaired mucosal barrier function, or "leaky gut" , which results in increased gut permeability, is caused by epithelial-damaging substances linked to industrialization, urbanization and modern life, such as household and dishwashing cleaning agents and the use of (ultra) processed foods through, amongst others, emulsifiers.

An intact mucosal barrier is crucial for the maintenance of tissue homeostasis as this protects against allergens. An increased gut permeability can result in an enhanced uptake of allergens where they may activate the immune system leading to severe chronic inflammation. Thus, it is well possible that an impaired mucosal barrier function may contribute to these observed differences in threshold to peanut and nuts.

Mucosal barrier dysfunction has been demonstrated in asthma, chronic rhinosinusitis, atopic dermatitis, and Eosinophilic Esophagitis (EoE) and a number of studies in food allergy. Both the Lactulose/Mannitol ratio in urine (L/M ratio) as well as the Raffinose/Mannitol ratio in urine (R/M ratio) are commonly used Sugar Absorption Tests (SAT) for the analysis of small intestinal permeability. In the Netherlands the R/M ratio has been implemented as sugar absorption test (SAT) and is provided by Good Manufacturing Practice (GMP) certified pharmacists. If the mucosal integrity is impaired the urinary excretion of Raffinose will increase (see methods for more details). In children, for example, increased gut permeability in milk- and egg allergic children was found as compared to 7 controls. Similar results were found by Andre et al in children and adults with sensitization to foods, 0,6 - 70 years. In a study in which the relationship between allergic symptoms and mucosal permeability was studied, a significant correlation between small intestine permeability and the severity of allergic symptoms at referral was shown.

The influence of nutrition on gut permeability:

Nutrition is one of the important external factors contributing to the maintenance of an intact mucosal barrier function of the gut. In contrast, unhealthy nutrition or nutrition containing barrier-damaging agents contributes to the disruption of the mucosal barrier through the following processes:

1. Direct effects of foods and nutrients on the maintenance or disruption of the mucosal integrity in the gut.

   Vitamin A plays a critical role in the differentiation of cells towards mucosal barrier function. Zinc and iron have an essential role in the maintenance of intestinal epithelial tight junction barrier via the regulation of claudin-3 and occluding expression. Short chain fatty acids produced through the microbial fermentation of dietary fiber, maintain mucosal integrity by processes including mucus production, tissue repair and up- regulation of the expression of tight junction proteins.

   In a small study in adult patients with eosinophilic esophagitis, it was shown that the intake of sunflower oil and/or stir fry oil, as well as the total amount of added fat, was negatively (i.e., unfavorably) related to in vitro values of permeability, while the consumption of buttermilk/yoghurt drink with Lactobacillus rhamnosus, dairy and vitamin A were favorably related to mucosal permeability of the esophagus.

   In contrast nutrition may also may have deleterious effects on the mucosal barrier function. Emulsifiers in highly processed foods are surfactants that behave like detergents, and even trace amounts of these agents markedly increase bacterial translocation in mouse models. Advanced Glycation End products (AGE) formation and additives commonly used by the food industry in highly processed foods play a role.

   Thus, our diet may be one of the key factors in the maintenance or impairment of our epithelial barrier function, and may as such contribute to the prevention and treatment of chronic immune disorders.
2. Our diet is an important source for the composition of our microbiome and regulation of the mucosal barrier function.

   Healthy dietary constituents feed our gut microbiota by providing substrates for a large variety of intestinal microbial species, leading to a diverse and anti-inflammatory microbiome. Dietary fiber, vegetables, legumes, grains, nuts, fish, plant-based foods, fermented dairy (e.g. buttermilk and yoghurt), omega-3 polyunsaturated fatty acids n-3 and polyphenols have anti-inflammatory capacity through modulation of our gut microbiota composition with a protective effect on our mucosal barrier function by regulation of tight junction barriers. Higher intake of animal foods, saturated fat, processed foods, alcohol and sugar induce pro-inflammatory processes by the reduction of the total abundance and reduction of specific species of bacteria in our gut and subsequent negative impact on our mucosal barrier function. Plant-based proteins and n-3 polyunsaturated fatty acids induce the opposite effect alongside increased abundance of anti-inflammatory species.
3. Nutrition provides nutrients which are essential for the functioning of the innate and adaptive immune system, which in turn regulate the mucosal barrier function. T cells, type 2 innate lymphoid cells (IL2) and interleukine 13 (IL13)play major roles. According to very strict criteria several nutrients are recognized by European Food Safety Authority (EFSA) for their immunomodulatory properties. These are copper, folate, iron, selenium, vitamin A, B6, B12, C, D and zinc.
4. Our diet can induce either pro-inflammatory or anti-inflammatory effects in the gut and our body. Diet is established among the most important influences on health in modern societies. Poor diet is among the leading causes of chronic disease. The composition of our diet may importantly enhance or reduce inflammation and may therefore influence inflammatory disease such as asthma and atopic dermatitis, This cannot be contributed to single foods, instead, the total dietary pattern is important. A Western diet which is characterized by a high consumption of meat, highly processed foods, ready-to-use foods and meals, refined grains, sugar, omega-6 fatty acids and saturated fatty acids, and a low consumption of dietary fiber, omega 3 fatty acids, anti-oxidants, fruits, vegetables and plant-based foods. Such a diet induces a pro-inflammatory state of our immune system and increased intestinal permeability.

In contrast, dietary patterns such as a traditional Mediterranean diet, with high contents of monounsaturated (MUFA), ω-3 polyunsaturated fatty acid, home-made meals, fruits, vegetables, legumes, and grains, has shown anti-inflammatory effects when compared with typical North American and Northern European dietary patterns. With regards to allergic disease specifically, the use of organic dairy and unprocessed milk is associated with lower prevalence of allergic diseases, as was shown in the KOALA birth cohort study and studies on children on farms.

Taken together, for peanut and nut allergy there is yet no cure and threshold levels to peanut or nuts differ widely for reasons unknown. Peanut and nut allergy often present in patients with coexisting atopic diseases such as atopic dermatitis and atopic asthma, which are based on inflammatory processes. An impaired mucosal barrier may contribute to the observed differences in thresholds to peanut and nuts. Nutrition can either positively or negatively influence our immune function, gut microbiota composition and gut permeability, and therefore may influence threshold levels to peanut and nuts, as well as severity of coexistent symptoms such as atopic dermatitis and asthma.

Thus, a study on dietary intervention as proposed in this protocol will yield lacking knowledge on the effect of a healthful diet on gut permeability and clinical symptoms in allergic disease.

The study will be performed in children as peanut and nut allergy are often lifelong, may be severe, cannot yet be cured and has a significant impact on quality of life which is underestimated by parents. The risk of inadvertent allergic reactions specifically holds for children with a low threshold to peanut. With a higher threshold level fewer products need to be avoided which will improve quality of life. In addition, comorbidity in allergic disease such as eczema is most prominent in children. Therefore, children will most benefit from our study results if we can show immune-supportive diet improves gut barrier function and alleviates allergic symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Children of 3 to 17 years of age with a positive open or double-blind placebo-controlled peanut or nut challenge < 12 months to inclusion OR an obvious and objective IgE-mediated allergic reaction following the consumption of isolated peanut or nut within 1 hours, confirmed by sensitisation to peanut or nut < 24 months to inclusion;
* Children who are potty trained or house trained;
* Presence of IgE to peanut ≥0.35 kilo units per liter (kU/l) or skin prick test > 3 mm to peanut or nut, < 12 months prior to challenge.

Exclusion Criteria:

* Only mild symptoms in the oral cavity to peanut or nut due to pollen food syndrome;
* A negative peanut or nut challenge;
* Children who are not potty trained (house trained);
* Gastro-intestinal diseases (e.g. Morbus Crohn, coeliac disease, Colitis Ulcerosa), lactose intolerance
* severe cow's milk allergy -because of possible traces of cow's milk in lactose in the SAT), syndromes, infectious/immunology diseases other than atopy, or diabetes;
* Laxative treatment, such as lactulose;
* Not able to read or write Dutch.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 132 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in small intestine permeability between baseline and after 4 months of dietary intervention as expressed by the Raffinose/Mannitol ratio in urine | 4 months
  We will measure the ratio of Raffinose/Mannitol in urine at baseline and after 4 months of dietary intervention

SECONDARY OUTCOMES:
Relationship between gut permeability and the severity of atopic dermatitis | At baseline
  Gut permeability is measured by R/M ratio. Severity of atopic dermatitis is measured by SCORAD
Relationship between gut permeability and patient reported outcomes of asthma and allergic rhinitis | At baseline
  Gut permeability is measured by R/M ratio. Severity of Asthma and allergic rhinitis symptoms are measured by the Onderzoek astma en hooikoorts bij kinderen questionnaire (Caratkids)
Relationship between gut permeability and patient reported outcomes of gastrointestinal symptoms | At baseline
  Gut permeability is measured by R/M ratio. Gastrointestinal symptoms are measured by the Birmingham irritable bowel syndrome (IBS) questionnaire in Dutch
Relationship between gut permeability and treshold levels to peanut or nuts | At baseline
  The relationship between gut permeability (R/M ratio) and threshold level to peanut or nuts established during the oral food challenge (cumulative mg peanut or nut protein);
Differences in gut microbiota composition | At baseline and after 4 months
  Microbiota compostion will be measured by by gene sequencing technology (16S methods)
Differences in severity of atopic dermatitis | At baseline and after 4 months
  Differences in severity of atopic dermatitis measured (Scorad-score)
Differences in atopic dermatitis (POEM) | At baseline and after 4 months
  Differences in atopic dermatitis (POEM)
Differences in asthma | At baseline and after 4 months
  Differences in asthma (Caratkids)
Differences in gastro-intestinal symptoms | At baseline and after 4 months
  Differences in gastro-intestinal symptoms (Birmingham IBS questionnaire, Dutch version)
Differences in use of medications | At baseline and after 4 months
  Use of medication will be registered by a Medication Registration Form (MRF).
Differences in upper respiratory tract infections (URTIs) | At baseline and after 4 months
  Differences in upper respiratory tract infections (URTIs) by questionnaire (numbe fo days, doctor's visits, antibiotics, days off from school or work
Differences in food allergy quality of Life | At baseline and after 4 months
  Food allergy quality of life will be measured by disease-specific and age-related quality of life questionnaires (FAQLQ-ChildForm, FAQLQ-ParentForm and FAQLQ-TeenagerForm)
Self-assessed dietary adherence and feasibility of the Immune-supportive diet (intervention group only) | 2,5 and 4 months
  Self-assessed dietary adherence and feasibility of the Immune-supportive diet (intervention group only) will be measured by Likert scales
Relationship between gut permeability and nutritional intake | At baseline and after 4 months
  Gut permeability is measured by R/M ratio Dietary intervention (in grams of food) will be assessed by three online 24-hour food recalls
Calcultated dietary adherence | At baseline and after 4 months
  Calculated dietary adherence by the researcher by the number of first and second choice foods in 3-days food diaries after 4 months of dietary intervention

CONTACTS AND LOCATIONS:
Locations (1):
- OLVG, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
As the database contains patient (coded) information the database can be shared under request